CLINICAL TRIAL: NCT07066111
Title: The Effect of Bupivacaine Liposome Preemptive Analgesia on Postoperative Pain and Delirium in Elderly Patients Undergoing Hip Fracture Surgery: A Randomized, Parallel Controlled Prospective Clinical Study
Brief Title: The Effect of Bupivacaine Liposome Preemptive Analgesia on Postoperative Pain and Delirium in Elderly Patients Undergoing Hip Fracture Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hongwei Shi, Director, Department of Anesthesia, Pain and Perioperative Medicine, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY 20250527-02
Record Dates: First submitted 2025-06-17; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Delirium
Keywords: preemptive analgesia; bupivacaine liposome; ip fracture surgery; postoperative delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Tramadol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intramuscularly (Placebo Comparator): The elderly patients with hip fractures who were randomly divided into the control group were injected tramadol 100mg intramuscularly.
  Interventions: Drug: Tramadol
- ultrasound-guided high iliofascial space block (Experimental): The elderly patients with hip fractures who were randomly divided into the experimental group were given ultrasound-guided high iliofascial space block
  Interventions: Drug: bupivacaine liposome (ultrasound-guided high iliofascial space block)

INTERVENTIONS:
Drug: Tramadol — The control group routinely injected tramadol 100mg(Tramal) intramuscularly
  Arms: intramuscularly
Drug: bupivacaine liposome (ultrasound-guided high iliofascial space block) — the experimental group was given ultrasound-guided high iliofascial space block: High-frequency linear probe (5-13 MHZ, Sonosite, USA) was used to identify the iliac bone, iliac muscle and deep circumiliac artery. Then a short oblique puncture needle was used, with the intraplanar technique, and the needle was inserted from the outside. When the needle tip reached the surface of the iliac muscle (iliac fascia space), 20ml of bupivacaine liposome was injected. After the operation, electrocardiogram monitoring(Mindray) was performed for 1 hour to observe adverse reactions.
  Arms: ultrasound-guided high iliofascial space block

SUMMARY:
To explore the effects of bupivacaine liposomes in preemptive analgesia for iliofascial block on postoperative pain and postoperative delirium in elderly patients with hip fractures, to optimize perioperative analgesia strategies, to reduce the incidence of postoperative delirium, and to improve patient prognosis.

DETAILED DESCRIPTION:
The incidence of hip fractures has risen significantly with population aging. In 2016, the incidence of hip fractures in China was 177 per 100,000 for women and 99 per 100,000 for men, and it is projected that the number of hip fracture surgeries worldwide will reach 6.3 million by 2050. Surgical treatment is preferred among elderly hip fracture patients, but postoperative delirium (POD) is a common complication, with an incidence rate of 4.0%-53.3%, which is much higher than that of elective surgery patients (3.6%-28.3%). POD is closely associated with increased morbidity, mortality and medical expenses, and its mechanism is complex, involving sleep disorders, acute traumatic stress and inflammatory responses.

Elderly people have underlying diseases such as decreased multi-system functions (for example, organ-specific or chronic diseases) and decreased sensory functions (for example, visual and hearing impairments), and hip fractures can cause pain and functional loss. Pain is A Class A risk factor for POD, and about 42 percent of elderly patients with hip fractures experience moderate to severe pain during the acute phase. Pain not only triggers the release of inflammatory factors but also reduces sleep quality, further increasing the risk of POD. Therefore, effective perioperative analgesia is crucial for reducing the incidence of POD.

Regional nerve block analgesia (such as iliofascial block, FIB) has been widely used in recent years because of its definite analgesic effect and few side effects. Bupivacaine liposomes, as a new type of long-acting local anesthetic, can achieve stable drug release within 72 hours after injection and provide long-acting analgesia, but its effect on POD is not yet clear. This study aims to explore the effect of bupivacaine liposomes on preemptive analgesia of iliofascial block on postoperative pain and POD in elderly patients with hip fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hip fractures scheduled for surgical treatment (including femoral neck fractures, intertrochanteric fractures, and fractures more than 5 cm below the lesser trochanter of the femur).
* Age ≥65 years.
* American Society of Anesthesiologists (ASA) grade I - III.
* The patient or family member signed the informed consent form

Exclusion Criteria:

* Compound injuries (such as combined fractures of the head, chest, pelvis, or limbs).
* Have a clear history of mental illness or are taking psychotropic drugs.
* Preoperative delirium or the use of delirium-related medications (such as olanzapine).
* A history of acute cerebrovascular disease (cerebral infarction or cerebral hemorrhage) within 6 months.
* Patients requiring sedation or postoperative coma due to the condition.
* Allergy to amide local anesthetics.
* Severe arrhythmia or liver or kidney dysfunction

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
POD incidence | Evaluated twice daily within 3 days after surgery (8:00-10:00 and 18:00-20:00)
  Evaluated via the CAM scale.
  * CAM diagnostic criteria:
    1. Acute onset of mental changes and fluctuating course of the disease.
    2. Inattentiveness.
    3. Disordered thinking.
    4. Changes in consciousness levels.
  * A POD is diagnosed if it meets 1+2 or 1+3 or 1+4.

SECONDARY OUTCOMES:
Preoperative pain | before the surgery.
  Evaluate rest and exercise pain via VAS score (0-10)and record the consumption of analgesics.The higher the VAS score, the more severe the pain will be.
Postoperative pain | twice a day for 1-3 days after the operation
  Evaluate rest and exercise pain via VAS score (0-10).
Number of participants with Sleep quality | from hospitalization to 3 days after surgery(22:30-06:30).
  Sleep quality monitored by Cardiopulmonary coupling instrument.The cardiopulmonary coupling (CPC) technology utilizes heart rate variability to measure the function of the autonomic nervous system, and combines it with the extracted respiratory signals from the electrocardiogram (ECG) to generate a sleep profile. Using the CPC device, data such as single-lead ECG signals, sleep duration, respiratory events, activity level, and body position of the patients during sleep are monitored for data analysis to evaluate their sleep conditions.
Recovery quality | 24 hours after surgery
  Evaluated by QoR-15 score.QoR-15 was used to assess five aspects of postoperative recovery quality (physical comfort, physical independence, psychological support, emotion and pain), with higher scores indicating the higher postoperative recovery quality. The lowest score is 0 points, and the highest score is 150 points.
Anesthesia method form | during operation
  Anesthesia method of the surgery
intraoperative medication checklist | during operation
  intraoperative medication of the surgery
Number of participants with hemodynamic changes | during the operation
  hemodynamic changes during the operation.The changes in blood pressure, heart rate, blood oxygen saturation,body temperature and EtCO2 of the patients during the surgery were recorded through the monitoring equipment provided by Mindray.
postoperative complications | Periprocedural
  postoperative complications after the surgery
length of hospital stay | Periprocedural
  length of hospital stay
30-day mortality | 30-day after surgery
  30-day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China